CLINICAL TRIAL: NCT04387617
Title: Effect of Cannabidiol Oil on Postoperative Pain After Ureteroscopy for Urinary Calculi
Brief Title: A Study to Assess the Effect of Cannabidiol Oil on Pain After Ureteroscopy for Kidney Stones
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Karen L. Stern, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 19-011832
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Results first posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-12

CONDITIONS: Urinary Stone
MeSH Terms: conditions — Urinary Calculi | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CBD Oil Group (Experimental)
  Interventions: Drug: Cannabidiol
- Control Group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — The product is a liquid formulation that will be prescribed at a dosage of 20 mg per day for a total of 3 days.
  Other Names: Epidiolex
  Arms: CBD Oil Group
Drug: Placebo — The product is a liquid formulation placebo that will be prescribed at an equivalent volume as active drug for 3 days
  Arms: Control Group

SUMMARY:
The purpose of this study is to determine if CBD oil has any effect on decreasing postoperative pain control following ureteroscopy for urinary stone disease, and to determine if CBD oil has any effect in decreasing the amount of postoperative opioids (commonly used drug) used by patients after undergoing ureteroscopy for urinary stone disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with kidney or ureteral stones confirmed on imaging (CT of the abdomen and pelvis) and who elect for definitive treatment via ureteroscopy at two sites within a tertiary care institution.
* Age 18-75 years of age.
* Patients of either gender.
* Patients of all ethnic backgrounds.
* Capable of giving informed consent.
* Capable and willing to fulfill the requirements of the study.

Exclusion Criteria:

* History of chronic pain.
* Chronic use of opioid or other pain medication (> 12 weeks).
* Known allergy to CBD oil or other cannabinoids.
* Known or suspected pregnancy.
* Inability to give informed consent or unable to meet requirements of the study for any reason.
* Bilateral ureteroscopy.
* Current marijuana, cannabidiol (CBD), or dronabinol use.
* Liver disease/cirrhosis.
* Current treatment of seizures with clobazam, valproate, or other antiepileptic medications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Stern, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- CBD Oil Group: Cannabidiol: The product is a liquid formulation that was prescribed at a dosage of 20 mg per day for a total of 3 days.
- Control Group: Placebo: The product is a liquid formulation placebo that was prescribed at an equivalent volume as active drug for 3 days
Period: Overall Study
Arm/Group | CBD Oil Group | Control Group
Started | 45 | 45
Completed | 45 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBD Oil Group | Control Group | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (12.3) | 58.0 (14.4) | 59.7 (13.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 55
  Male | 17 | 18 | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Maximum Pain Intensity Score
Description: Patient self-reported maximum pain intensity score measured by the Visual Analogue Scale (VAS) rated from 0-10, where 0 was no pain and 10 was the worst pain imaginable.
Time Frame: postoperative Day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBD Oil Group | Control Group
Number analyzed (Participants) | 45 | 45
score on a scale | 3.6 (2.4) | 3.2 (2.8)
Statistical Analysis 1: Comparison: CBD Oil Group vs Control Group; Test type: Superiority; p = 0.5, t-test, 2 sided; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.8 to 1.6], Standard Deviation 2.6

2. Secondary Outcome: Postoperative Rescue Narcotic Use
Description: The number of subjects who required rescue narcotic use post ureteroscopy
Time Frame: postoperative Day 3
Measure: Count of Participants; unit: Participants
Arm/Group | CBD Oil Group | Control Group
Number analyzed (Participants) | 45 | 45
Participants | 8 | 9

3. Secondary Outcome: Total Urinary Symptoms Score
Description: Patient self-reported urinary symptoms measured by the Ureteric Stent Symptoms Questionnaire (USSQ) urinary symptoms section. Following insertion of the stents, subjects were asked to answer 11 questions regarding their urinary symptoms. 9 questions used a score of 1 to 5, where 1 was never and 5 was all of the time. 1 question used a score of 1 to 4, where 1 was do not see any blood and 4 was urine is heavily blood stained. 1 question used a score of 1 to 7, where 1 was delighted and 7 was terrible. Total sum of all 11 questions for a total score ranging from 11 - 56, lower scores reflected fewer symptoms and higher satisfaction where higher scores reflected more symptoms and less satisfaction.
Time Frame: postoperative day 1 and postoperative day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBD Oil Group | Control Group
Number analyzed (Participants) | 45 | 45
score on a scale
  Postoperative day 1 | 31 (5.5) | 33 (6.6)
  Postoperative day 3 | 27 (5.8) | 27 (6.9)

4. Secondary Outcome: The Number of Subjects With Adverse Events
Description: The count of subjects who experienced adverse events
Time Frame: 3 days post-ureteroscopy
Measure: Count of Participants; unit: Participants
Arm/Group | CBD Oil Group | Control Group
Number analyzed (Participants) | 45 | 45
Participants
  Nausea | 3 | 2
  Constipation | 10 | 9
  Diarrhea | 3 | 1
  Poor appetite | 8 | 4
  Poor sleep | 11 | 5
  Drowiness | 11 | 8
  Dizziness | 7 | 5
  Tiredness | 17 | 13
  Itching | 2 | 2
  Headache | 4 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected from each subject from baseline to end of study for a total of 3 days
Arm/Group | CBD Oil Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 24/45 | 21/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CBD Oil Group (N=45) | Control Group (N=45)
Nausea (General disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 10 | 9
Diarrhea (Gastrointestinal disorders) | 3 | 1
Poor Appetite (Metabolism and nutrition disorders) | 8 | 4
Poor sleep (Psychiatric disorders) | 11 | 5
Drowsiness (Nervous system disorders) | 11 | 8
Dizziness (Nervous system disorders) | 7 | 5
Tiredness (General disorders) | 17 | 13
Itching (Skin and subcutaneous tissue disorders) | 2 | 2
Headache (Nervous system disorders) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT04387617/Prot_SAP_000.pdf